CLINICAL TRIAL: NCT05427890
Title: Evaluation of Diabetes Risk Communication Tool to Promote Behaviour Change for Prevention of Type 2 Diabetes
Brief Title: Diabetes Risk Communication Tool Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Principal Investigator, Huso Yi, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OF-LCG-RiskComm; NUS-IRB-2021-633 (Other: National University, Singapore)
Record Dates: First submitted 2022-06-10; First posted 2022-06-22 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator)
  Interventions: Behavioral: T2D Risk Communication Tool: Traffic Light
- Relative Risk (Experimental)
  Interventions: Behavioral: T2D Risk Communication Tool: Relative Risk
- Metabolic Age (Experimental)
  Interventions: Behavioral: T2D Risk Communication Tool: Metabolic Age

INTERVENTIONS:
Behavioral: T2D Risk Communication Tool: Relative Risk — Risk of T2D is presented in comparison to the rest of the Singapore population in a scale 1-10. Suggestions on different lifestyle changes and its potential to reduce the individual's relative risk is presented for user to observe impact of preventative behaviours.
  Arms: Relative Risk
Behavioral: T2D Risk Communication Tool: Metabolic Age — Risk of T2D is presented as an age, compared to their chronological age as a proxy for their current health status. Suggestions on different lifestyle changes and its potential to reduce the individual's metabolic age is presented for user to observe impact of preventative behaviours.
  Arms: Metabolic Age
Behavioral: T2D Risk Communication Tool: Traffic Light — Risk of T2D is presented as either High (Red) or Low (Green). Generic tips on how to reduce risk of diabetes are included. This imitates the tool that is currently available for residents of Singapore to use to assess their risk of T2D.
  Arms: Usual Care

SUMMARY:
Prevention for Type 2 Diabetes (T2D)has been vast but with limited success. While Singaporeans have high knowledge about T2D, its symptoms, and risk factors, healthy practices are still sub-optimal. Upon a qualitative investigation, it was found that there is little to no urgency to engage in T2D preventative behaviour due to to the low perceived threat, and high costs from required lifestyle changes relative to the benefits. Hence, this project targets to communicate the risk of diabetes in a more salient and effective way to improve the intention of preventative behaviour by targeting the constructs of Protection Motivation Theory (PMT) and increasing the threat and coping appraisals. The current available diabetes risk assessment tool's result page provides a binary output: "Higher vs Lower" Risk of being pre-diabetic. This aligns with the usual care practiced in clinics currently; patients are told if they are pre-diabetic or not. It does not provide any personalized or relevant tips on how to reduce risk. Hence, there was a demonstrated need to develop risk assessment tools that increase threat appraisal and communicate T2D risk in a more salient way to motivate the intention of behaviour change. The investigators developed two tools: Relative Risk, and Metabolic Age. The Relative Risk prototype demonstrates the user's relative risk on a scale of 1 to 10, in comparison to someone of the same age and sex. The number 1-10 represents their position in the percentile distribution of their risk scores. The Metabolic Age is identified by matching the risk score's percentile position to percentile of the incidence of T2D. The median age of the people in that percentile is reflected as the metabolic age. The primary objectives of this study is to evaluate which of these risk presentations (Usual care, relative risk, or metabolic age) evoke (i) effective cognitive and emotional responses to risk results and (2) motivation for the intention of behaviour change. The secondary objective is to provide empirical evidence for using PMT constructs in intervention development. The hypothesis is that those who are exposed to the Metabolic Age risk assessment and communication tool will have the most effective cognitive and emotional response, and the highest intention of engaging in behaviour change, followed by those exposed to relative risk, and then standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-60 years;
* Singapore citizen, or permanent resident
* Able to read and understand English,
* Have had a health screening with blood pressure, triglycerides, and HbA1C done within the last 3 months
* At least one risk factor for Type 2 Diabetes (BMI ≥ 23 kg/m2, blood pressure ≥130/85 mmHg or receiving therapy for hypertension, triglycerides ≥1.7mmol/L or HbA1c ≥5.7%)

Exclusion Criteria:

- Diagnosis of any event of cardiovascular disease, kidney issues, or type 2 diabetes

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 460 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Differences in reaction to risk communication between arms | 1 day
  Participants' emotional responses to their risk results are assessed using 6 items like "I found the results worrying" and "I am reassured by these results". 3 additional items are used to assess their reaction to the process and confidence towards the tool by asking about their understanding of the results and if they will encourage others to use the tool. Participants will answer these on a 5-point scale, ranging from 'strongly disagree' to 'strongly agree.'
  Participants' cognitive reactions to their risk results are assessed using 3 items to evaluate their risk perception in five years, ten years, and in relation to others. Participants will answer these on a 5-point scale, ranging from 'very unlikely' to 'very likely.'
Differences in behaviour intention between arms | 1 day
  Assessed using 10 items to understand the intention to improve their health-promoting behaviours after they have gone through one of the risk assessment tools. Items ask questions like "After seeing my results, I intend to have fewer sugary drinks (soda, fruit juice, bubble tea) in a week" and "After seeing my results, I intend to do more moderate to vigorous exercise (ie brisk walking, jogging, weight lifting, etc) in a week" Responses are evaluated on a 5-point scale, from "Extremely Unlikely to Extremely Likely".

SECONDARY OUTCOMES:
Empirical evidence of using PMT constructs in developing interventions | 1 day
  We measure the different PMT constructs (perceived severity, perceived vulnerability, response efficacy, self-efficacy, and response costs). This will allow us to observe how the different tools differ and if these constructs are associated with the primary outcome measures. Responses are evaluated on a 7-point scale, ranging from 'definitely disagree' to 'definitely agree.'

OTHER OUTCOMES:
Objective Risk Score | 1 day
  We collect the health screening data the participants are using to engage with the risk assessment tools to compute their objective risk scores. This will allow us to observe any associations between the different risk groups (ie low, moderate, or high) and the primary and secondary outcome measures. Data used in the risk model to calculate the objective risk score: age, sex, height, weight, systolic and diastolic blood pressure, use of blood pressure medication, triglycerides, HbA1C, parental history of T2D, and average exercise minutes per week.

CONTACTS AND LOCATIONS:
Overall Officials: Huso Yi, PhD, Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore